CLINICAL TRIAL: NCT01657058
Title: The Effects of Different Modes of Administration of Soluble Fibre on Postprandial and Second Meal Blood Glucose Response, Appetite and Sensory Parameters in Healthy Individuals
Brief Title: Effects of Mode of Administration of Soluble Fibre Blend on Glycemia, Appetite & Sensory Parameters
Acronym: FI-FORM
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Unity Health Toronto (Other)
Responsible Party: Principal Investigator, Vladimir Vuksan, Professor, Unity Health Toronto
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 12-147
Record Dates: First submitted 2012-08-01; First posted 2012-08-03 (Estimated); Last update posted 2014-03-07 (Estimated); Status verified 2014-03

CONDITIONS: Healthy
Keywords: soluble fiber; second meal effect; glycemia; satiety; Individuals

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (5):
- Treatment # 1 (Experimental): Soluble viscous fibre blend powder in hydrophobic matrix
  Interventions: Dietary Supplement: Soluble viscous fibre blend powder in hydrophobic matrix
- Treatment # 2 (Experimental): Soluble viscous fibre blend in pre hydrated form
  Interventions: Dietary Supplement: Soluble viscous fibre blend in pre hydrated form
- Control # 1 (Placebo Comparator): No soluble viscous fibre blend
  Interventions: Dietary Supplement: No soluble viscous fibre blend
- Treatment # 3 (Experimental): Soluble viscous fibre blend premixed with ½ carbohydrate gel
  Interventions: Dietary Supplement: Soluble viscous fibre blend premixed with ½ carbohydrate gel
- Control # 2 (Placebo Comparator): No soluble viscous fibre blend, ½ carbohydrate jello
  Interventions: Dietary Supplement: No soluble viscous fibre blend, ½ carbohydrate jello

INTERVENTIONS:
Dietary Supplement: Soluble viscous fibre blend powder in hydrophobic matrix — 5g soluble viscous fibre blend pre-mixed into margarine (hydrophobic matrix) + white bread + jello
  Arms: Treatment # 1
Dietary Supplement: Soluble viscous fibre blend in pre hydrated form — 0g soluble viscous fibre blend margarine + white bread +5g Konjac fibre prehydrated in jello
  Arms: Treatment # 2
Dietary Supplement: No soluble viscous fibre blend — 0g soluble viscous fibre blend margarine + white bread + jello
  Arms: Control # 1
Dietary Supplement: Soluble viscous fibre blend premixed with ½ carbohydrate gel — Margarine + white bread (1/2 carbohydrate) +5g soluble viscous fibre blend hydrated in jello with glucose
  Arms: Treatment # 3
Dietary Supplement: No soluble viscous fibre blend, ½ carbohydrate jello — Margarine + white bread (1/2 carbohydrate) +5g soluble viscous fibre blend hydrated in jello with glucose
  Arms: Control # 2

SUMMARY:
Soluble, viscous fibre has been established as an effective dietary component for lowering postprandial glycemia and promoting satiety. The effectiveness of viscous fibre has been related to its ability to increase the viscosity of the intra-luminal contents of the small intestine. Hence, the proposed mechanism with which soluble fibre affects the glycemic response, dependent on the viscosity development in the gut, would require that soluble fibre be extractable from the food matrix. This, in part, may be dependent on the food matrix that the soluble fibre is incorporated in. While properties of soluble fibre and their physiological effects have been studied extensively, limited data exists on the most effective mode of administration of fibre to optimize benefits. Furthermore, there are no studies to date that have evaluated how different modes of highly viscous soluble fibre would affect the subsequent meal. Hence, we propose a research study to determine whether the form of administration, taking into consideration the carbohydrate availability of a viscous fibre blend supplement, has a significant impact on postprandial and second meal glycemic response and subjective satiety in healthy individuals.

DETAILED DESCRIPTION:
Following a 10-12 hr overnight fast, subjects will visit the Risk Factor Modification Centre between 8:00 am and 1:00 pm. Blood pressure and anthropometric measurements, including body weight, height, and % body fat will be taken. An initial finger prick fasting blood sample will be taken and a subjective appetite questionnaire in the form of a 100 mm visual analog scale will be completed. Subsequently, one of the 5 study meals will be administered to the subject to consume over a 10-15 minute duration accompanied by 300ml of water. Subjects will then be asked to complete a palatability questionnaire. Over the following 3 hours capillary blood samples will be taken by finger pricks at 15, 30, 45, 60, 90, 120 and 180 minutes post treatment. Appetite and symptoms questionnaires will be completed at 15, 30, 45, 60, 75, 90, and 120. At 180 min, a second standardized meal will be administered, consisting of 400kcal of pizza and 200ml of water. Further finger pick blood samples will be taken at 15, 30, 45, 60 and 120 min post pizza consumption. Upon completion of the visit, subjects will be given a 24-hour symptoms questionnaire to complete at home as an additional safety measure for a 24-hour period.

ELIGIBILITY:
Inclusion Criteria:

* age 18-65 years
* normal glycemic response
* BMI between 18.5 - 25 kg/m2
* peripheral systolic and diastolic blood pressure <140 mmHg and <90 mmHg, respectively.

Exclusion Criteria:

* Known reported history of liver or kidney disease, diabetes, hypertension, stroke or myocardial infarctions, thyroid disease, Celiac disease/gastrointestinal disease, or AIDS
* allergies to any of the test products
* Presence of an eating disorder
* Following a restrictive dieting regime
* Weight loss of >5kg in last 2 months
* Smoking cigarettes
* Alcohol intake >2 drinks/day
* using prescription medications or Natural Health Products;
* any condition which, in the opinion of the investigator might jeopardize the health and safety of the subject or study personnel, or adversely affect the study results

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2012-07; Primary Completion 2012-12 (Actual); Study Completion 2014-10 (Estimated)

PRIMARY OUTCOMES:
Postprandial glycemia | 5 hours
  To investigate the effectiveness of soluble dietary fibre blend supplementation depending on 1) mode of administration and 2) carbohydrate incorporation on reducing postprandial glycemia when consumed with a standardized test breakfast.

SECONDARY OUTCOMES:
Satiety | 5 hours
  To investigate the effectiveness of soluble dietary fibre blend supplementation depending on 1) mode of administration and 2) carbohydrate incorporation on subjective satiety when consumed with a standardized test breakfast.
  At each visit, participants will record their subjective ratings using a 100mm visual analogue scale and these ratings will be combined into a total subjective appetite score.
Second Meal Glycemia | 2 hours
  To investigate the effectiveness of these different methods of administration of konjac fibre blend on postprandial glycemia of the second standardized meal.
Palatability | 5 hours
  At each visit, participants will record their subjective ratings using a 100mm visual analogue scale and these ratings will be combined into a total subjective palatability score.

CONTACTS AND LOCATIONS:
Overall Officials: Vladimir Vuksan, Principal Investigator — Unity Health Toronto
Locations (1):
- St.Michael's Hospital, Toronto, Ontario, Canada